CLINICAL TRIAL: NCT01107769
Title: A Single-center, Randomized, Value Study of VISIONAIRE™ Patient Matched Technology vs. Standard Surgical Instrumentation
Brief Title: VISIONAIRE™ Value Study
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VISVAL01
Record Dates: First submitted 2010-04-09; First posted 2010-04-21 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VISIONAIRE™: Total knee arthroplasty with VISIONAIRE™ patient-matched cutting blocks
- Standard Instrumentation: Total knee arthroplasty with standard instrumentation

SUMMARY:
This is a single center randomized observational study that evaluates the cost benefit ratio between the use of two types of instrumentation in TKA: standard instrumentation vs. VISIONAIRE™ Patient Matched Technology. This study does not involve treatment or investigational products, as all components are FDA approved and are commercially available.

DETAILED DESCRIPTION:
The objective of the current observational study is to assess value of surgical instrumentation following analysis of health economic data. It is hypothesized that patient matched cutting block technology VISIONAIRE™ may reduce TKA operative time, blood loss, surgical error and adverse event risk as well as providing improved mechanical alignment. In order to test this hypothesis, subjects will be randomized to either VISIONAIRE™ or standard TKA instrumentation groups. One site will enroll a total of 38 patients; 19 patients per group. All patients meeting the inclusion/exclusion criteria specified in this protocol will be asked to participate in the study. If the patient consents to participate, they will be enrolled in the study and randomized to one of the two study arms. Patients requiring TKA will be implanted with Legion, Genesis II or Journey BCS (Smith & Nephew) total knee implant systems. Standard instrumentation will be used to assist the surgeon in placing the implant in the control group. In the VISIONAIRE™ group, standard instrumentation will not be used in the surgery. Patients randomized to the VISIONAIRE™ arm will have an MRI preoperatively that will be used to create the customized cutting blocks. All patients will have an x-ray at each postoperative interval.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the inclusion criteria.

1. Patient is diagnosed with degenerative joint disease of the knee requiring a unilateral TKA.
2. Patient is of legal age to consent, and is skeletally mature.
3. Patient is willing to sign and date an IRB/IEC approved consent form.

Exclusion Criteria:

Patients must not meet any of the exclusion criteria.

1. Patient has poor bone stock making a TKA unjustifiable.
2. Patient has active, local infection or previous intra-articular infections.
3. Patient has neuropathic (Charcot) joint.
4. Patient is pregnant or may become pregnant during the course of the study.
5. Patient is severely overweight (BMI >40).
6. Patient is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population considered for this study includes patients with osteoarthritis (degenerative joint disease)of the knee requiring unilateral TKA.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Health Economic Criteria | Up to 6 weeks
  This study will evaluate the cost benefit ratio between the use of two types of instrumentation in TKA: standard instrumentation vs. VISIONAIRE™. The following will be collected & reported from the OR and discharge report:
  * instrument tray set-up time
  * operative time
  * blood loss
  * instrumentation requirements
  * discharge disposition
  * ambulatory support on discharge
  * adverse event

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a measure of Safety and Tolerability | Perioperative & Postoperative (up to 6 weeks)
  Radiographic analysis will be conducted to assess preoperative and postoperative mechanical alignment between groups. All perioperative and postoperative surgical or instrument-related adverse events will be recorded during this study.

CONTACTS AND LOCATIONS:
Overall Officials: John Noble, Jr, M.D., Principal Investigator — Center for Orthopaedics Lake Charles, LA
Locations (1):
- John Noble, Jr., Lake Charles, Louisiana, United States

REFERENCES:
- [Result] J Arthroplasty. 2011 Sep 9. [Epub ahead of print] http://www.ncbi.nlm.nih.gov/pubmed/21908169
- [Result] Noble JW Jr, Moore CA, Liu N. The value of patient-matched instrumentation in total knee arthroplasty. J Arthroplasty. 2012 Jan;27(1):153-5. doi: 10.1016/j.arth.2011.07.006. Epub 2011 Sep 9. PMID 21908169
- See also: The Value of Patient-Matched Instrumentation in Total Knee Arthroplasty. — http://www.ncbi.nlm.nih.gov/pubmed/21908169